CLINICAL TRIAL: NCT06245902
Title: A Clinical Trial to Assess a Single Dose of Low-Dose Naltrexone and Acetaminophen Combination and Its Components in the Acute Treatment of Migraine
Brief Title: An Acute Migraine Factorial Study
Acronym: ANODYNE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allodynic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANODYNE-1 Version 1.3
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Migraine With or Without Aura
Keywords: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Naltrexone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Factorial Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Naltrexone and Acetaminophen (Experimental): Patients take one capsule containing naltrexone and one capsule containing acetaminophen together for a qualifying migraine
  Interventions: Drug: Naltrexone and Acetaminophen
- Naltrexon/Acetaminophen-High Capsules (Experimental): Patient take one capsule containing naltrexone (high dose) and one capsule containing acetaminophen together for a qualifying migraine
  Interventions: Drug: Naltrexone and Acetaminophen-High Dose
- Naltrexone Alone Capsules (Active Comparator): Patient take one capsule containing naltrexone and one capsule containing placebo together for a qualifying migraine
  Interventions: Drug: Naltrexone Alone (regular dose)
- Acetaminophen Alone Capsules (Active Comparator): Patient take one capsule containing naltrexone and one capsule containing placebo together for a qualifying migraine
  Interventions: Drug: Acetaminophen Alone
- Placebo Capsules (Placebo Comparator): Patient take two capsule containing placebo together for a qualifying migraine
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Naltrexone and Acetaminophen — Naltrexone plus acetaminophen
  Arms: Naltrexone and Acetaminophen
Drug: Naltrexone and Acetaminophen-High Dose — Naltrexon (high dose) plus acetaminophen
  Arms: Naltrexon/Acetaminophen-High Capsules
Drug: Naltrexone Alone (regular dose) — Naltrexone Alone plus Placebo
  Arms: Naltrexone Alone Capsules
Drug: Acetaminophen Alone — Acetaminophen Alone plus Placebo
  Arms: Acetaminophen Alone Capsules
Drug: Matching Placebo — Two Placebo capsules
  Arms: Placebo Capsules

SUMMARY:
The study consists of a screening visit, out-patient treatment of a moderate or severe migraine attack with a single dose of the study medication within 8 weeks, and End-of-Study Visit 2-7 days after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. History of migraine with or without aura according to the International Classification of Headache Disorders (ICHD)-3rd edition (beta version) for at least one-year with first migraine prior to age 50.
3. Migraine-associated nausea with ≥half of migraine attacks.
4. 2 - 8 migraines per month in each of the previous 3 months.
5. The patient is able to complete study questionnaires, comply with the study requirements and restrictions, and willing to provide written informed consent and authorize HIPAA.
6. The female patient who is premenopausal or postmenopausal less than 1 year, or have not had surgical sterilization (i.e., tubal ligation, partial or complete hysterectomy) must have a negative urine pregnancy test, be non-lactating, and commit to using adequate and reliable contraception throughout the study (e.g., barrier with additional spermicidal, intra-uterine device, hormonal contraception). The male patient must be surgically sterile or commit to the use of 2 different methods of birth control during the study and for 28 days after taking the study drug.

Exclusion Criteria:

1. The patient in the opinion of the investigator, may have medication-overuse headache pain (as defined by ICHD - 3 beta criteria for medication-overuse headache), (analgesic, opioid, ergotamine or triptan overuse) during the 3 months preceding screening.
2. The patient in the opinion of the investigator has chronic migraine (as defined by ICHD - 3 beta criteria for chronic migraine).
3. History of cluster headache or neurologically complicated migraine (hemiplegic, basilar, retinal, ophthalmoplegic migraine).
4. Initiation or change in medications with possible migraine prophylactic effects during 3 months before inclusion into the trial (E.g., calcium channel blockers, tricyclic antidepressants, beta-blockers, selective serotonin re-uptake inhibitors (SSRIs), serotonin-norepinephrine re-uptake inhibitors (SNRIs), or Botox).
5. Any concurrent medical or psychiatric condition, this includes, but is not limited to chronic unstable debilitating diseases, significant renal or hepatic impairment.
6. A history within the previous 3 years of abuse of any drug, prescription, illicit, or alcohol.
7. The Female patient is pregnant or breast-feeding. The Male patient is not practicing 2 different methods of birth control with their partner during the study, and for 28 days after the investigational drug last dose or will not remain abstinent during the study, and for 28 days after the last dose.
8. Use of opiates or barbiturates more than 3 days per month.
9. Known-hypersensitivity reaction to any of the components of the investigational drug.
10. Consumption of analgesic medication for other conditions on a regular basis, (nonsteroidal anti-inflammatory drugs, or acetaminophen, or muscle relaxants).
11. Use of emergency care treatment more than 3 times in the previous 6 months.
12. Participation in another study with an investigational drug within 30 days prior to randomization and/or a plan to participate during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
% of patients reporting no headache pain. | 2 hours post-dose
  Self-reported headache pain on a four-point Likert scale.
% of patients having absence of most bothersome migraine-associated symptom (MBS). | 2 hours post-dose
  MBS was prospectively identified at baseline. Self-reported MBS as present or absent.
% of patients who have "sustained pain freedom" | 24-hour post-dose.
  Defined as having no headache pain at 2 hours after dose, with no use of rescue medication and no relapse of headache pain within 24 hours after administration of the investigational drug.

SECONDARY OUTCOMES:
% of patients having absence of nausea, photophobia, phonophobia, and neck/shoulder pain | 24-hour post-dose.
  Self-reported the current status of their associated symptom as present or absent.
% of patients who used rescue medications | 2-24 hours
% of patients who had headache pain relapse. | 2-48 hours
  Defined as the return of headache of any severity within 48 hours after administration of the investigational drug, when the patient was pain-free at 2 hours after the administration of the investigational drug.

OTHER OUTCOMES:
% of patients who experienced adverse events | 48 hours
  treatment related Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Annette C Toledano, M.D., Study Director — Allodynic Therapeutics, Inc
Locations (1):
- Annette C. Toledano MD, North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Zhang Y, Peng Y, Hutchinson MR, Rice KC, Yin H, Watkins LR. Pharmacological characterization of the opioid inactive isomers (+)-naltrexone and (+)-naloxone as antagonists of toll-like receptor 4. Br J Pharmacol. 2016 Mar;173(5):856-69. doi: 10.1111/bph.13394. Epub 2016 Feb 4. PMID 26603732
- [Result] Kato J, Svensson CI. Role of extracellular damage-associated molecular pattern molecules (DAMPs) as mediators of persistent pain. Prog Mol Biol Transl Sci. 2015;131:251-79. doi: 10.1016/bs.pmbts.2014.11.014. Epub 2015 Jan 30. PMID 25744676
- [Result] Lewis SS, Loram LC, Hutchinson MR, Li CM, Zhang Y, Maier SF, Huang Y, Rice KC, Watkins LR. (+)-naloxone, an opioid-inactive toll-like receptor 4 signaling inhibitor, reverses multiple models of chronic neuropathic pain in rats. J Pain. 2012 May;13(5):498-506. doi: 10.1016/j.jpain.2012.02.005. Epub 2012 Apr 20. PMID 22520687
- [Result] Watkins LR, Hutchinson MR, Ledeboer A, Wieseler-Frank J, Milligan ED, Maier SF. Norman Cousins Lecture. Glia as the "bad guys": implications for improving clinical pain control and the clinical utility of opioids. Brain Behav Immun. 2007 Feb;21(2):131-46. doi: 10.1016/j.bbi.2006.10.011. Epub 2006 Dec 18. PMID 17175134
- [Result] Hutchinson MR, Zhang Y, Brown K, Coats BD, Shridhar M, Sholar PW, Patel SJ, Crysdale NY, Harrison JA, Maier SF, Rice KC, Watkins LR. Non-stereoselective reversal of neuropathic pain by naloxone and naltrexone: involvement of toll-like receptor 4 (TLR4). Eur J Neurosci. 2008 Jul;28(1):20-9. doi: 10.1111/j.1460-9568.2008.06321.x. PMID 18662331
- [Result] Wieseler J, Ellis A, McFadden A, Stone K, Brown K, Cady S, Bastos LF, Sprunger D, Rezvani N, Johnson K, Rice KC, Maier SF, Watkins LR. Supradural inflammatory soup in awake and freely moving rats induces facial allodynia that is blocked by putative immune modulators. Brain Res. 2017 Jun 1;1664:87-94. doi: 10.1016/j.brainres.2017.03.011. Epub 2017 Mar 16. PMID 28322750
- [Result] Su M, Ran Y, He Z, Zhang M, Hu G, Tang W, Zhao D, Yu S. Inhibition of toll-like receptor 4 alleviates hyperalgesia induced by acute dural inflammation in experimental migraine. Mol Pain. 2018 Jan-Dec;14:1744806918754612. doi: 10.1177/1744806918754612. Epub 2018 Jan 8. PMID 29310498
- [Result] Dewall CN, Macdonald G, Webster GD, Masten CL, Baumeister RF, Powell C, Combs D, Schurtz DR, Stillman TF, Tice DM, Eisenberger NI. Acetaminophen reduces social pain: behavioral and neural evidence. Psychol Sci. 2010 Jul;21(7):931-7. doi: 10.1177/0956797610374741. Epub 2010 Jun 14. PMID 20548058
- [Result] Younger J, Mackey S. Fibromyalgia symptoms are reduced by low-dose naltrexone: a pilot study. Pain Med. 2009 May-Jun;10(4):663-72. doi: 10.1111/j.1526-4637.2009.00613.x. Epub 2009 Apr 22. PMID 19453963
- [Result] Lipton RB, Baggish JS, Stewart WF, Codispoti JR, Fu M. Efficacy and safety of acetaminophen in the treatment of migraine: results of a randomized, double-blind, placebo-controlled, population-based study. Arch Intern Med. 2000 Dec 11-25;160(22):3486-92. doi: 10.1001/archinte.160.22.3486. PMID 11112243
- [Result] Kaki AM, El-Yaski AZ, Youseif E. Identifying neuropathic pain among patients with chronic low-back pain: use of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):422-8. doi: 10.1016/j.rapm.2005.05.013. PMID 16135345
- See also: 2009-2013 Pain Research Advances | Interagency Pain ...Thus, identifying potential new medications is critical. Recent evidence indicates a pivotal role for the receptor known as toll-like receptor 4 (TLR4 ... — https://search.usa.gov/search?utf8=%E2%9C%93&affiliate=iprcc&query=tlr4&x=0&y=0